CLINICAL TRIAL: NCT01255020
Title: Safety and Efficacy Evaluation of Restricted Protein Dietary Supplemented With α-keto Acid on Protecting Residual Renal Function in CAPD Patients--A Prospective, Double Blind Randomized, Parallel Control, Multi-center Clinical Trial
Brief Title: Renal Protective Effects of Restricted Protein Dietary With α-keto Acid in CAPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Beijing Fresenius Kabi Pharmaceutical Co (Industry)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KAPDRRF
Record Dates: First submitted 2010-08-11; First posted 2010-12-07 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Renal Function Disorder
Keywords: α-Keto Acid; Restricted Protein Diet; Residual Renal Function
MeSH Terms: interventions — Diet, Protein-Restricted; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- α-Keto Acid plus restricted protein diet (Active Comparator): Participants randomized to this group will receive 12 months treatment of α-Keto Acid. The dose of α-Keto Acid is 100mg/kg per day and will divided into three times per day, and the α-Keto Acid will be asked to be taken during the meal. In addition, the participants will be asked to restrict the protein intake. The protein intake is restricted as 1g/kg/d.
  Interventions: Drug: α-Keto Acid with restricted protein diet
- Placebo plus restricted protein diet (Placebo Comparator): All participants will receive 12 months treatment of placebo, at the same time they will be asked to restrict the protein intake.The dose of placebo is 100mg/kg per day, and the protein intake is restricted as 1g/kg/d.
  Interventions: Drug: Placebo plus restricted protein diet

INTERVENTIONS:
Drug: α-Keto Acid with restricted protein diet — α-Keto Acid: The daily dose of compound α-Keto Acid is 100mg/kg/d. The total daily dose will be divided into three times a day.
  Restricted Protein Diet: Diet contain protein 1.0g/kg/d
  Other Names: Test Group
  Arms: α-Keto Acid plus restricted protein diet
Drug: Placebo plus restricted protein diet — placebo: The daily dose of placebo is 100mg/kg/d. The total daily dose will be divided into three times a day.
  Diet contain protein 1.0 g/kg/d.
  Other Names: Control Group
  Arms: Placebo plus restricted protein diet

SUMMARY:
The prospective, double blind randomized, parallel control, and multi-center clinical trial will evaluate the safety and efficacy of α-keto acid with restricted protein diet on protecting residual renal function in continuous ambulatory peritoneal dialysis (CAPD) patients.

DETAILED DESCRIPTION:
Residual renal function (RRF) is associated with cardiovascular complication, nutritional status, incidence of peritonitis, and quality of life in peritoneal dialysis (PD) patients. Therefore, RRF is an important determinant of mortality and morbidity in PD patients.

Previous studies have suggested that dietary protein restriction supplemented with α-keto acids may slow the loss of RRF in chronic kidney disease patients. However, these trials are small sample and short-time research. In PD patients, there is very few reports to indicate the effect of α-keto acid with restricted protein diet on RRF.

The aim of this study is to evaluate the safety and efficacy of α-keto acid with restricted protein diet on protecting residual renal function in continuous ambulatory peritoneal dialysis (CAPD) patients.This is a prospective, double blind randomized, parallel control, and multi-center clinical study. 160 patients who meet Inclusion/Exclusion criteria will be randomized into α-Keto Acid group or control group at the ratio of 1:1. The α-Keto Acid group will use compound α-Keto Acid plus restricted protein diet, while control group will use placebo plus restricted protein diet.The α-Keto Acid dosage is 100mg/kg/d daily. The restricted protein dosage is 1g/kg/d. The safety and efficacy of α-Keto Acid with restricted protein diet on RRF will be evaluated after 1 year treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients on peritoneal dialysis (PD) at least three month prior to study entry.
2. Subjects of either sex, more than 18 years old, the range of age is 18 to 70 year old.
3. Residual GFR ≥ 3 ml/min/1.73m2.
4. Without α-Keto Acid therapy in recent 4 weeks.
5. Subjects who agree to participate in the study and sign the informed consent.

Exclusion Criteria:

1. History of peritonitis or other infection within one month.
2. Patients with insufficient dialysis.
3. History of taking drug which may influence amino acid metabolism within one month(glucocorticoid, thyroxin, antithyroid drug, androgens,amino acids,et al).
4. Patients with diseases which contraindicate ketosteril.
5. Cannot control diet according to protocol.
6. Alcohol abuse or drug abuse.
7. Having malignant tumor.
8. History of psychiatric or neuropathic dysfunction.
9. Cardiac failure, with New York Heart Association (NYHA) grade III-IV or history of severe heart and cerebrovascular disease in recent one month(acute stroke, acute heart failure, Lability angina)
10. Serum albumin < 30g/l.
11. Serum calcium > 2.8mmol/l.
12. Participation in another clinic trial within last three months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The longitudinal change in residual glomerular filtration rate (GFR) | Every 3 months up to 12 months

SECONDARY OUTCOMES:
Peritoneal membrane transport characteristics | Every 3 months up to 12 months
Cardiovascular events | Every 3 months up to 12 months
Nutritional status | Every 3 months up to 12 months
Hospitalization | Every 3 months up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing YU, M.D. & Ph.D., Principal Investigator — 1st Affiliated Hospital, Sun Yat-Sen University; Lan Chen, M.D. & Ph.D, Principal Investigator — Ruijin Hospital; Jianghua Chen, M.D. & Ph.D, Principal Investigator — First Affiliated Hospital of Zhejiang University; Zhangsuo Liu, M.D. & Ph.D, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Fei Xiong, M.D., Principal Investigator — Wuhan Chinese and Western Medicine Combined Hospital; Qinfeng Han, M.D.&Ph.D, Principal Investigator — Peking University Third Hospital
Locations (1):
- The 1st Affiliated Hospital, Sun Yet-sen University, Guangzhou, Guangdong, China